CLINICAL TRIAL: NCT05163028
Title: A Phase 1, Open-Label, Dose Escalation of HBI-2376 in Patients With Advanced Malignant Solid Tumors Harboring KRAS or EGFR Mutations
Brief Title: A Dose Escalation Study of SHP2 Inhibitor in Patients With Solid Tumors Harboring KRAS of EGFR Mutations
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBI-2376-101
Record Dates: First submitted 2021-11-24; First posted 2021-12-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer; Colorectal Cancer; Pancreatic Cancer; Solid Tumor; Cancer; Cancer of Pancreas; Cancer of Colon
Keywords: KRAS; EGFR; SHP2; FIH
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 Dose Escalation Design with Expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): HBI-2376 will be given orally in ascending doses (escalation cohort), until the maximum tolerated dose or recommended Phase 2 dose is reached. Up to 6 patients will then be enrolled in the expansion cohort at the recommended dose.
  Interventions: Drug: HBI-2376

INTERVENTIONS:
Drug: HBI-2376 — SHP2 Inhibitor

SUMMARY:
A Phase 1 dose escalation study in patients with advanced solid tumors harboring KRAS or EGFR mutations to determine the maximum tolerated dose and recommended Phase II dose of HBI-2376 and characterize its pharmacokinetic profile.

DETAILED DESCRIPTION:
A Phase 1, Open-Label, Dose Escalation of HBI-2376 in Patients with Advanced Malignant Solid Tumors Harboring KRAS or EGFR Mutations. The primary and secondary objectives are:

1. To determine the MTD and recommended Phase 2 dose (RP2D), of HBI-2376 as an oral monotherapy for advanced solid tumors harboring KRAS or EGFR mutations
2. To characterize the PK of HBI-2376 in subjects with advanced malignant solid tumors harboring KRAS or EGFR mutations

HBI-2376 is a SHP2 Inhibitor and will be dosed once daily throughout the escalation and expansion phase. Up to 42 subjects will be enrolled sequentially into the 3+3 dose escalation and monitored throughout the study for safety and tolerability. The dose escalation phase will consist of 6 cohorts, with doses ranging from 6 to 40mg. Once the MTD of RP2D is established, additional 6 subjects will be enrolled into the expansion phase at that dose level.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female at least 18 years of age at the time of signing the ICF prior to initiation of any study specific activities/procedures
* Advanced malignant solid tumors with KRAS or EGFR mutations diagnosed by histology or cytology
* Relapsed or refractory to, or intolerant of, or refuse approved or standard of care established therapy known to provide clinical benefit for disease
* At least 1 measurable target lesion that meets the definition of RECIST v1.1
* ECOG Performance Status of 0 or 1
* Demonstrate adequate organ function
* Must be able to swallow oral medications and must not have gastrointestinal abnormalities that significantly affect drug absorption

Key Exclusion Criteria:

* History of another concurrent malignancy within 3 years prior to study entry, unless the malignancy was treated with curative intent and the likelihood of relapse is <5% in 2 years Note: Subjects with a history of squamous or basal cell carcinoma of the skin or carcinoma in the situ of the cervix may be enrolled
* Untreated or symptomatic central nervous system (CNS) metastases Note: Subjects with asymptomatic treated CNS metastases are eligible provided they have been clinically stable and not requiring steroids for at least 4 weeks
* Clinically significant cardiovascular disease, including stroke or myocardial infarction within 6 months
* Any unresolved Grade 2 or greater toxicity from previous anti-cancer therapy, except alopecia, within 4 weeks of first study treatment administration
* Active autoimmune diseases or history of autoimmune diseases that may relapse
* Pregnant or nursing
* Prior treatment with any SHP2 inhibitors
* Any condition that required systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤14 days before the first study treatment administration
* Treatment with other investigational drugs/devices within 4 weeks prior to first study treatment administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D), of HBI-2376 as an oral monotherapy for advanced solid tumors harboring KRAS or EGFR mutations. | Up to 36 months
  Safety endpoints: Incidence of dose-limiting toxicities (DLTs), adverse events (AEs), and serious adverse events (SAEs) overall, by severity, by relationship to HBI-2376, and those that led to discontinuation of HBI-2376

SECONDARY OUTCOMES:
Pharmacokinetic variables including maximum plasma concentration (Cmax) | Cycle 1 (28 days)
  Pharmacokinetic variables including maximum plasma concentration (Cmax)
Pharmacokinetic variables including minimum plasma concentration (Cmin) | Cycle 1 (28 days)
  Pharmacokinetic variables including minimum plasma concentration (Cmin)
Pharmacokinetic variables including Area Under the Curve (AUC) | Cycle 1 (28 days)
  Pharmacokinetic variables including Area Under the Curve (AUC)
Pharmacokinetic variables including clearance | Cycle 1 (28 days)
  Pharmacokinetic variables including clearance
Pharmacokinetic variables including serum half-life | Cycle 1 (28 days)
  Pharmacokinetic variables including serum half-life
Pharmacokinetic variables including volume of distribution | Cycle 1 (28 days)
  Pharmacokinetic variables including volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Salgia, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (12):
- United States (11):
  - City of Hope, Duarte, California
  - California Cancer Associates for Research and Excellence, Inc. (cCare), Encinitas, California
  - Providence Medical Foundation, Fullerton, California
  - California Cancer Associates for Research and Excellence, Inc. (cCare), San Marcos, California
  - Sarcoma Oncology, Santa Monica, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - Orlando Health, Inc., Orlando, Florida
  - BRCR Medical Center, Plantation, Florida
  - Gabrail Cancer Center, Canton, Ohio
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Pan American Center for Oncology Trials (PanOncology Trials), Rio Piedras, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: No